CLINICAL TRIAL: NCT05678361
Title: Sleep's Influence on the Treatment of Intrusive Emotional Memories With Trauma-focused CBT
Brief Title: Sleep's Influence on the Treatment of Intrusive Emotional
Acronym: SLEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-01357
Record Dates: First submitted 2018-09-17; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Intrusive Memories; PTSD
Keywords: sleep; memory; consolidation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Psychotherapists and outcome assessors are blind to participants' group membership (i.e., sleep versus wake after exposure therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep after exposure (Experimental): Participants take a nap during 90 min following three exposure (WET) sessions.
  Interventions: Behavioral: Sleep/Nap
- Wake after exposure (No Intervention): Participants watch a 90 min documentary following three exposure (WET) sessions.

INTERVENTIONS:
Behavioral: Sleep/Nap — Participants sleep after a maximum of three sessions of exposure therapy.
  Arms: Sleep after exposure

SUMMARY:
Intrusive memories represent a debilitating core feature of PTSD, one of the most prevalent psychiatric disorders following trauma. Exposure therapy is amongst the most successful treatments of PTSD that is recommended by most of the current national and international guidelines. The current study aims to test whether sleep as adjunct to written exposure sessions, a type of exposure- based treatment for PTSD, may boost the effectiveness of the therapy.

DETAILED DESCRIPTION:
Intrusive memories represent a debilitating core feature of PTSD, one of the most prevalent psychiatric disorders following trauma. Exposure therapy is amongst the most successful treatments of PTSD that is recommended by most of the current national and international guidelines. However, not all patients benefit equally and only about 50% show sustained response. There is thus room for improvement in terms of (i) better understanding who benefits from this type of therapy and (ii) possible ways of augmenting existing trauma-focused therapies. The current study aims to contribute to these endevours. Specifically, the study aims to test whether sleep as adjunct to written exposure sessions, a type of exposure- based treatment for PTSD, may boost the effectiveness of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* DSM V criteria of PTSD (at least moderate symptoms in two categories)
* Currently receiving Written Exposure Therapy at one of the psychotherapy centers at the Psychiatric University Clinic (PUC).
* Not more than moderate alcohol consumption (not more than 5 alcoholic drinks/week).
* Ability to understand the study instructions

Exclusion Criteria:

* Travel over > 3 time zones in < 3 months
* head injury
* shift work
* current substance abuse
* neurological disease
* drug addiction
* Current suicidality

Specific exclusion criteria for the fMRI:

* Acute psychotic symptoms
* Pregnancy
* Claustrophobia
* Magnetic resonance imaging incompatibility:
* Cardiac pacemaker or other metallic implants (e.g. metallic cardiac valve, insulin pump)
* Metallic foreign particles (e.g. after bullet wound, shell splinter, clips, metal prostheses)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Clinician- assessed Posttraumatic stress symptom severity at 1 week | One week post- treatment
  Clinician- assessed PTSD symptom severity (CAPS- 5)
Self-reported Posttraumatic stress symptom severity at 1 week | One week post- treatment
  Self - reported PTSD symptom severity (PCL-5)
Clinician- assessed Posttraumatic stress symptom severity at 1 month | One month post- treatment
  Clinician- assessed PTSD symptom severity (CAPS- 5)
Self-reported Posttraumatic stress symptom severity at 1 month | One month post- treatment
  Self - reported PTSD symptom severity (PCL-5)

SECONDARY OUTCOMES:
Total sleep time | Immediately after written exposure therapy
  Total sleep time according to EEG
Time spent in N1 sleep | Immediately after written exposure therapy
  N1 time according to EEG
Time spent in N2 sleep | Immediately after written exposure therapy
  N2 time according to EEG
Time spent in N3 sleep | Immediately after written exposure therapy
  N3 time according to EEG

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Kleim, PhD, Principal Investigator — Zurich
Locations (1):
- Psychiatric University Hospital, Zurich, Canton of Zurich, Switzerland